CLINICAL TRIAL: NCT00002575
Title: A PHASE III PROSPECTIVE RANDOMIZED TRIAL COMPARING LAPAROSCOPIC-ASSISTED COLECTOMY VERSUS OPEN COLECTOMY FOR COLON CANCER
Brief Title: Laparoscopic-Assisted Surgery Compared With Open Surgery in Treating Patients With Colon Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-934653; NCI-2012-02234 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CAN-NCIC-CO12; CDR0000063648 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-04-10 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer
Keywords: stage I colon cancer; stage II colon cancer; stage III colon cancer; adenocarcinoma of the colon
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional surgery (Experimental): Patients undergo open laparotomy and colectomy. A standard incision is made through the abdominal wall and the abdominal cavity is explored. A right or left colectomy or a sigmoid resection is performed.
  Patients may be entered on adjuvant chemotherapy trials after surgery provided the subsequent trial does not include radiotherapy and allows entry of patients from both arms.
  Quality of life is assessed at baseline and on days 2 and 14 after surgery, at 2 months, and then at 18 months. (closed as of 4/30/99)
  Patients are followed every 3 months for 1 year, every 6 months for 4 years, and then annually for 3 years.
  Interventions: Procedure: conventional surgery
- Laparoscopic-assisted colectomy (Experimental): Patients undergo a laparoscopic-assisted colectomy. A small infraumbilical incision is made through the abdominal skin and the abdominal cavity is insufflated with CO2 to allow access and visualization. The abdominal cavity is explored. If advanced local disease is identified, a celiotomy and colectomy are performed. Otherwise, a right or left colectomy or sigmoid resection is performed using laparoscopic-assisted techniques.
  Patients may be entered on adjuvant chemotherapy trials after surgery provided the subsequent trial does not include radiotherapy and allows entry of patients from both arms.
  Quality of life is assessed at baseline and on days 2 and 14 after surgery, at 2 months, and then at 18 months. (closed as of 4/30/99)
  Patients are followed every 3 months for 1 year, every 6 months for 4 years, and then annually for 3 years.
  Interventions: Procedure: laparoscopic surgery

INTERVENTIONS:
Procedure: conventional surgery
  Arms: Conventional surgery
Procedure: laparoscopic surgery
  Arms: Laparoscopic-assisted colectomy

SUMMARY:
RATIONALE: Less invasive types of surgery may help reduce the number of side effects and improve recovery. It is not yet known which type of surgery is more effective for colon cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of laparoscopic-assisted colectomy with open colectomy in treating patients who have colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the disease-free and overall survival rates of patients with colon cancer treated with laparoscopic-assisted colectomy vs open colectomy.
* Compare the safety of these regimens in terms of early and late morbidity and 30-day mortality of these patients.
* Compare the differences in costs and cost effectiveness between these treatments in this patient population.
* Compare the differences in quality of life of patients treated with these regimens. (closed as of 4/30/99)

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, primary surgeon, site of primary tumor (right vs left vs sigmoid), and American Society of Anesthesiologists disease classification (I and II vs III). Patients are randomized to one of two treatment arms.

The extent of colon resection is identical for both arms.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Clinical diagnosis of primary adenocarcinoma

  * Involving a single colon segment:

    * Right colon from the ileocecal valve up to and including the hepatic flexure
    * Left colon from the splenic flexure to the junction of the sigmoid and descending colon
    * Sigmoid colon between the descending colon and the rectum (at least 15 cm from the dentate)
* Diagnosis based on physical exam plus either a proctosigmoidoscopy and barium enema or a colonoscopy
* No advanced local disease that renders laparoscopic resection impossible
* No acutely obstructed or perforated colon cancer requiring urgent surgery
* No transverse colon cancer (i.e., between distal hepatic flexure and proximal splenic flexure)
* No stage IV disease
* No rectal cancer (i.e., below the peritoneal reflection, lower edge of tumor less than 15 cm from dentate)
* No American Society of Anesthesiologists IV/V disease classification
* No associated gastrointestinal diseases (i.e., Crohn's, chronic ulcerative colitis, or familial polyposis) that require additional extensive operative evaluation or intervention

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Other:

* No other prior or concurrent malignancy within the past 5 years except superficial squamous cell or basal cell skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Surgery:

* No prohibitive scars/adhesions from prior abdominal surgery

Other:

* No concurrent investigational treatments or invasive diagnostic procedures within 30 days after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 810 (Actual)
Dates: Start 1994-08; Primary Completion 2004-05 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | Up to 8 years
  * Compare the disease-free and overall survival rates of patients with colon cancer treated with laparoscopic-assisted colectomy vs open colectomy.
  * Compare the safety of these regimens in terms of early and late morbidity and 30-day mortality of these patients.
  * Compare the differences in costs and cost effectiveness between these treatments in this patient population.
  * Compare the differences in quality of life of patients treated with these regimens. (closed as of 4/30/99)
Overall survival | Up to 8 years

SECONDARY OUTCOMES:
Morbidity | Up to 8 years
Mortality | At 30 days
Costs and cost effectiveness between these treatments in this patient population | Up to 8 years
Compare the differences in quality of life of patients treated with these regimens | Up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Nelson, MD, Study Chair — Mayo Clinic
Locations (158):
- United States (145):
  - Huntsville Hospital System, Huntsville, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - St. Mary's Hospital, Rogers, Arkansas
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - Scripps Clinic, La Jolla, California
  - University of California San Diego Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Saint Mary Medical Center - Long Beach, Long Beach, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Naval Medical Center - Oakland, Oakland, California
  - Sutter Cancer Center, Sacramento, California
  - Veterans Affairs Satellite Clinic - Sacramento, Sacramento, California
  - Naval Medical Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Baptist Regional Cancer Institute - Jacksonville, Jacksonville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical College of Georgia Comprehensive Cancer Center, Augusta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - MBCCOP-Cook County Hospital, Chicago, Illinois
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Illinois Masonic Medical Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - West Suburban Hospital Medical Center, Oak Park, Illinois
  - Rockford Clinic, Rockford, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Regional Cancer Center, Indianapolis, Indiana
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Lucille Parker Markey Cancer Center, University of Kentucky, Lexington, Kentucky
  - Norton Healthcare System, Louisville, Kentucky
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Louisiana State University Medical Center - New Orleans, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Franklin Square Hospital Center, Baltimore, Maryland
  - National Naval Medical Center, Bethesda, Maryland
  - Regional Cancer Therapy Center - Frederick, Frederick, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Clinic - Burlington, Burlington, Massachusetts
  - Berkshire Medical Center, Pittsfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Memorial Healthcare, Worester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - St. Louis University School of Medicine, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Cancer Center - Omaha, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of New Mexico Cancer Research & Treatment Center, Albuquerque, New Mexico
  - Albany Regional Cancer Center, Albany, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Genesee Surgical Associates, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Akron City Hospital, Akron, Ohio
  - Aultman Cancer Center, Canton, Ohio
  - Jewish Hospital of Cincinnati, Inc., Cincinnati, Ohio
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - South Pointe Hospital, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - Oregon Cancer Center, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Network - Bethlehem, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Kent County Memorial Hospital, Warwick, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Baptist Regional Cancer Center - Knoxville, Knoxville, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Medical Group of Texas, Dallas, Texas
  - Kelsey Seybold Clinic, Houston, Texas
  - Wilford Hall - 59th Medical Wing, Lackland Air Force Base, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Texas Health Center at Tyler, Tyler, Texas
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Vermont Cancer Center, Burlington, Vermont
  - Virginia Oncology Associates - Newport News, Newport News, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - CCOP - Green Bay, Green Bay, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (11):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Royal Victoria Hospital - Montreal, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital - Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - L'Hopital Laval, Ste-Foy, Quebec
- Puerto Rico (2):
  - MBCCOP - San Juan, San Juan
  - Veterans Affairs Medical Center - San Juan, San Juan

REFERENCES:
- [Result] Stucky CC, Pockaj BA, Novotny PJ, Sloan JA, Sargent DJ, O'Connell MJ, Beart RW, Skibber JM, Nelson H, Weeks JC. Long-term follow-up and individual item analysis of quality of life assessments related to laparoscopic-assisted colectomy in the COST trial 93-46-53 (INT 0146). Ann Surg Oncol. 2011 Sep;18(9):2422-31. doi: 10.1245/s10434-011-1650-2. Epub 2011 Mar 31. PMID 21452066
- [Result] Larson DW, Marcello PW, Larach SW, Wexner SD, Park A, Marks J, Senagore AJ, Thorson AG, Young-Fadok TM, Green E, Sargent DJ, Nelson H. Surgeon volume does not predict outcomes in the setting of technical credentialing: results from a randomized trial in colon cancer. Ann Surg. 2008 Nov;248(5):746-50. doi: 10.1097/SLA.0b013e31818a157d. PMID 18948801
- [Result] Clinical Outcomes of Surgical Therapy Study Group; Nelson H, Sargent DJ, Wieand HS, Fleshman J, Anvari M, Stryker SJ, Beart RW Jr, Hellinger M, Flanagan R Jr, Peters W, Ota D. A comparison of laparoscopically assisted and open colectomy for colon cancer. N Engl J Med. 2004 May 13;350(20):2050-9. doi: 10.1056/NEJMoa032651. PMID 15141043
- [Result] Weeks JC, Nelson H, Gelber S, Sargent D, Schroeder G; Clinical Outcomes of Surgical Therapy (COST) Study Group. Short-term quality-of-life outcomes following laparoscopic-assisted colectomy vs open colectomy for colon cancer: a randomized trial. JAMA. 2002 Jan 16;287(3):321-8. doi: 10.1001/jama.287.3.321. PMID 11790211